CLINICAL TRIAL: NCT02828306
Title: Computer Based Algorithm for Patient Specific Implants for Cranioplasty in Patients With Skull Defects: a Prospective Clinical Trial
Brief Title: Computer Based Algorithm for Patient Specific Implants for Cranioplasty in Patients With Skull Defects
Acronym: CAPSID
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: CAPSID
Record Dates: First submitted 2016-06-21; First posted 2016-07-11 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Stroke; Head Trauma
Keywords: stroke; head trauma; Patient Specific Implant; skull defect
MeSH Terms: conditions — Stroke; Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with skull defects: Patients with skull defects after craniotomy for example tumor resection, head trauma, stroke which need a Patient Specific Implant.
  Interventions: Other: Patient Specific Implant

INTERVENTIONS:
Other: Patient Specific Implant — Implantation of Patient Specific Implant

SUMMARY:
Patients with skull defects after craniotomy for example tumor resection, head trauma, stroke, need a reimplantation of the bone afterwards. For some circumstances, their own bone cannot be reimplanted due to infection, tumor infiltration, damage to the bone, or aseptic bone necrosis. In these cases a Patient Specific Implant (PSI) needs to be designed to fit into the patient's skull defect.

The design of the PSI is based on the preoperative CT-scan of the patient's head with the skull defect, the imaging data set is uploaded and processed with IPlanNet software by BrainLab®. With the help of the software, a 3D model of a negative mould of the PSI is designed and printed. In the operation room, the PSI is fabricated under sterile conditions using the PSI mould. The design of the PSI mould with the help of IPlanNet is demanding and takes some few hours depending on the complexity of the case to be designed. In certain cases the accuracy of the fabricated PSI mould is not optimal, so that the surgeon intraoperatively has to adapt for the inaccuracy to achieve the best cosmetic and functional results at the expense of the operation duration, a known risk factor for postoperative wound infection and other perioperative complications.

Therefore, the investigators have developed an automated computer-based algorithm for PSI design (CAPSID). With the help of this tool, an accurate PSI and its corresponding mould can be calculated and designed based on the preoperative CT scan of the patient within 5-15 minutes and the corresponding mould can be printed. This step is automated and thus, independent of the neurosurgeons experience and skills in 3D processing software. The mould can be used for intraoperative fabrication of the implant under sterile conditions in the common way as described above. The possible advantages of the clinical establishment of this procedure would be a higher accuracy of the PSI compared to the conventional PSI fabrication method with better cosmetic results, lower costs and faster availability and production leading to shorter waiting time for the patient, and as a consequence of the higher accuracy leading to shorter operation time, with a reduction of risk of operative adverse events for the patient. Furthermore, the proof of practicability of this new method, could lead to new concepts in the field of Computer-based Patient Specific Implants in modern medicine in general.

DETAILED DESCRIPTION:
Patients with skull defects after craniotomy for example tumor resection, head trauma, stroke, need a reimplantation of the bone afterwards. For some circumstances, their own bone cannot be reimplanted due to infection, tumor infiltration, damage to the bone, or aseptic bone necrosis. In these cases a Patient Specific Implant (PSI) needs to be designed to fit into the patient's skull defect. Several materials are currently used such as titanium, poly-ether-ether-ketone (PEEK) or poly-methylmethyl-acrylate (PMMA) for PSI fabrication. At the moment, PSI are commercially available from different companies (DePuy Synthes®, EOS®, Xilloc®). Apart from the high costs of commercially available PSI, it takes usually several weeks until the designed and manufactured PSI is delivered to the hospital ready for reimplantation.

On the other hand, a method for software-based PSI design and intraoperative fabrication of the PSI under sterile conditions was described by Stieglitz et al. This method is currently used in everyday clinics in the department of neurosurgery in Bern. In short summary, the design of the PSI is based on the preoperative CT-scan of the patient's head with the skull defect, the imaging data set is uploaded and processed with IPlanNet software by BrainLab®. With the help of the software, a 3D model of a negative mould of the PSI is designed and printed. In the operation room, the PSI is fabricated under sterile conditions using the PSI mould. The design of the PSI mould with the help of IPlanNet is demanding and takes some few hours depending on the complexity of the case to be designed. In certain cases the accuracy of the fabricated PSI mould is not optimal, so that the surgeon intraoperatively has to adapt for the inaccuracy to achieve the best cosmetic and functional results at the expense of the operation duration, a known risk factor for postoperative wound infection and other perioperative complications.

Therefore, the investigators have developed an automated computer-based algorithm for PSI design (CAPSID). With the help of this tool, an accurate PSI and its corresponding mould can be calculated and designed based on the preoperative CT scan of the patient within 5-15 minutes and the corresponding mould can be printed. This step is automated and thus, independent of the neurosurgeons experience and skills in 3D processing software. The mould can be used for intraoperative fabrication of the implant under sterile conditions in the common way as described above. The possible advantages of the clinical establishment of this procedure would be a higher accuracy of the PSI compared to the conventional PSI fabrication method with better cosmetic results, lower costs and faster availability and production leading to shorter waiting time for the patient, and as a consequence of the higher accuracy leading to shorter operation time, with a reduction of risk of operative adverse events for the patient. Furthermore, the proof of practicability of this new method, could lead to new concepts in the field of Computer-based Patient Specific Implants in modern medicine in general. A clinical trial is necessary to proof the advantages and practicability of the investigators' concept of computer-based algorithm for PSI design (CAPSID) for patients with skull defects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with skull defects due to craniotomy who need a Patient Specific Implant (PSI) of the skull
* Age older than 18 and less than 90 years
* Provided written informed consent

Exclusion Criteria:

* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to Palacos
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the study
* Known coagulopathy
* Severe disease with limited life expectancy of less than one year

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with skull defects after craniotomy for example tumor resection, head trauma, stroke, need a Patient Specific Implant (PSI).
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2016-09; Primary Completion 2019-06 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Number of patients where there is no need to adapt the PSI's edges | 6 weeks after surgery by standardised questionnaire
Number of patients where there is no need to augment/fill clefts between the PSI and patient´s bone | 6 weeks after surgery by standardised questionnaire
Number of patients where there is no need to discard the PSI and fabricate a new PSI | 6 weeks after surgery by standardised questionnaire

SECONDARY OUTCOMES:
Operation duration | intraoperative
Patient's satisfaction measured by questionary | 6 weeks
infection rate | day 1-3 after OP, at 6 weeks
postoperative haemorrhage | day 1-3 after OP, at 6 weeks
postoperative cerebrospinal fluid leakage | day 1-3 after OP, at 6 weeks
PSI-displacement | day 1-3 after OP, at 6 weeks
need for reoperation | day 1-3 after OP, at 6 weeks
Accuracy of the PSI determined by volumetric analysis of the patient´s post-implantation CT scan (dice similarity index) | 3 days after surgery
Accuracy of the PSI determined by volumetric analysis of the patient´s post-implantation CT scan (volumetric inaccuracy index) | 3 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Schucht, MD, Principal Investigator — University Hospital Inselspital
Locations (1):
- Dep. of Neurosurgery, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Della Puppa A, Rustemi O, Gioffre G, Troncon I, Lombardi G, Rolma G, Sergi M, Munari M, Cecchin D, Gardiman MP, Scienza R. Predictive value of intraoperative 5-aminolevulinic acid-induced fluorescence for detecting bone invasion in meningioma surgery. J Neurosurg. 2014 Apr;120(4):840-5. doi: 10.3171/2013.12.JNS131642. Epub 2014 Jan 10. PMID 24410157
- [Background] Lassen B, Helseth E, Ronning P, Scheie D, Johannesen TB, Maehlen J, Langmoen IA, Meling TR. Surgical mortality at 30 days and complications leading to recraniotomy in 2630 consecutive craniotomies for intracranial tumors. Neurosurgery. 2011 May;68(5):1259-68; discussion 1268-9. doi: 10.1227/NEU.0b013e31820c0441. PMID 21273920
- [Background] Stieglitz LH, Fung C, Murek M, Fichtner J, Raabe A, Beck J. What happens to the bone flap? Long-term outcome after reimplantation of cryoconserved bone flaps in a consecutive series of 92 patients. Acta Neurochir (Wien). 2015 Feb;157(2):275-80. doi: 10.1007/s00701-014-2310-7. Epub 2014 Dec 24. PMID 25534126
- [Background] Chim H, Gosain AK. Biomaterials in craniofacial surgery: experimental studies and clinical application. J Craniofac Surg. 2009 Jan;20(1):29-33. doi: 10.1097/SCS.0b013e318190dd9e. PMID 19164984
- [Background] Stieglitz LH, Gerber N, Schmid T, Mordasini P, Fichtner J, Fung C, Murek M, Weber S, Raabe A, Beck J. Intraoperative fabrication of patient-specific moulded implants for skull reconstruction: single-centre experience of 28 cases. Acta Neurochir (Wien). 2014 Apr;156(4):793-803. doi: 10.1007/s00701-013-1977-5. Epub 2014 Jan 18. PMID 24442601